CLINICAL TRIAL: NCT04405037
Title: A Prospective Randomized Control Trial of The Effectiveness of Alvimopan as a Rescue Treatment of Postoperative Ileus Following Colorectal Surgery
Brief Title: Alvimopan as a Rescue Treatment of Postoperative Ileus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scott Steele (Other)
Responsible Party: Sponsor-Investigator, Scott Steele, Principle Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-321
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Ileus; Gastrointestinal Dysfunction
MeSH Terms: conditions — Ileus | interventions — alvimopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alvimopan Group (Experimental): Patients randomized to the study group will be given a maximum of 3 doses of Alvimopan 12mg orally, 12 hours apart. Alvimopan will be given from the time of diagnosis of postoperative ileus to the time of return of bowel function or the maximum 3 doses. Subsequent Alvimopan doses will be given if there is no return of bowel function or if symptoms of distension and/or nausea persist despite some return of bowel function.
  All patients will follow a standard ERAS pathway after surgery, with early feeding and ambulation, along with opioid minimizing measures as is our standard postoperative protocol.
  Interventions: Drug: Alvimopan
- Control Group (No Intervention): Control patients will follow a standard ERAS pathway after surgery, including NPO status, IV fluid rehydration, and nasogastric decompression, early feeding and ambulation, along with opioid minimizing measures as is our standard postoperative protocol.

INTERVENTIONS:
Drug: Alvimopan — Alvimopan will be given to patients who are diagnosed with postoperative ileus after surgery
  Other Names: Entereg
  Arms: Alvimopan Group

SUMMARY:
This study aims to evaluate the cost effectiveness of Alvimopan as rescue therapy in patients undergoing colorectal or small bowel resection who develop POI, and its safety and effectiveness in reducing LOS and POI duration.

This will be a prospective randomized control trial with a total of 58 patients, 29 in each group. Patients who undergo laparoscopic or open colorectal resection, small bowel resection, or ileostomy reversal with small bowel resection that subsequently develop postoperative ileus will be eligible for enrollment. If they meet inclusion/exclusion criteria, they will be randomized at the time of diagnosis of postoperative ileus to receive Alvimopan as rescue therapy or to receive conservative standard care.

Patients randomized to the study group will be given a maximum of 3 doses of Alvimopan 12mg orally, 12 hours apart. Alvimopan will be given from the time of diagnosis of postoperative ileus to the time of return of bowel function or the maximum 3 doses. Subsequent Alvimopan doses will be given if there is no return of bowel function or if symptoms of distension and/or nausea persist despite some return of bowel function.

DETAILED DESCRIPTION:
This study aims to evaluate the cost effectiveness of Alvimopan as rescue therapy in patients undergoing colorectal or small bowel resection who develop POI, and its safety and effectiveness in reducing LOS and POI duration.

Hypothesis:

The investigators hypothesize that the use of alvimopan as rescue therapy in patients undergoing colorectal and small bowel resection surgery who develop POI can shorten their duration of POI and hospital length of stay.

Objectives:

To perform a prospective RCT to evaluate the effect of alvimopan as rescue therapy compared to standard of care in reducing the duration of post-operative ileus and post-operative LOS after colorectal and small bowel resection surgery.

Protocol:

This will be a prospective randomized control trial with a total of 58 patients, 29 in each group. Patients who undergo laparoscopic or open colorectal resection, small bowel resection, or ileostomy reversal with small bowel resection that subsequently develop postoperative ileus will be eligible for enrollment. If they meet inclusion/exclusion criteria, they will be randomized at the time of diagnosis of postoperative ileus to receive Alvimopan as rescue therapy or to receive conservative standard care.

At the time of diagnosis of postoperative ileus and after enrollment and randomization, all patients will be returned to NPO status. Nasogastric tubes (NGT) may be placed for gastric decompression at the discretion of the surgical team if clinically indicated. In the event that an NGT is placed, medications will be given orally or via the NGT, which will be clamped for 30 minutes after administration. Patients will continue on standard ERAS pathways with the exception of reduction of diet. Antiemetics will be given as clinically indicated; however, no prokinetic or promotility agents will be given as scheduled dosages.

Patients randomized to the study group will be given a maximum of 3 doses of Alvimopan 12mg orally, 12 hours apart. Alvimopan will be given from the time of diagnosis of postoperative ileus to the time of return of bowel function or the maximum 3 doses. Subsequent Alvimopan doses will be given if there is no return of bowel function or if symptoms of distension and/or nausea persist despite some return of bowel function.

All patients will follow a standard ERAS pathway after surgery, with early feeding and ambulation, along with opioid minimizing measures as is our standard postoperative protocol.

The patient and surgical team will be able to know which arm of the study the patient is in based on documentation in the medical record of the administration of Alvimopan.

Standard discharge criteria will be applied to all patients, including: Passage of stool, Ability to tolerate solid food and to drink comfortably, Adequate oral analgesia, Patient's willingness to be discharged.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who have benign or malignant colonic or rectal disease that have undergone laparoscopic or open colorectal resection, small bowel resection or ileostomy reversal with small bowel resection and subsequently developed postoperative ileus, defined as:

  a. Patients with symptoms of bloating with or without nausea and vomiting, with absence of passage of flatus or stool who require either

  i. Return to NPO status after initial diet attempts

ii. Undergo placement of a nasogastric tube

b. Patients with absence of passage of flatus or stool who are either

i. More than 5 days after open surgery without recovery of GI function

ii. More than 3 days after laparoscopic surgery or ileostomy closure without recovery of GI function

2. Subjects who are 18 years of age and older

3. Subjects of either gender

4. Subjects who are willing and able to adhere to protocol requirements, agree to participate in the study program and provide written and informed consent.

Exclusion Criteria:

* 1. Subjects who received Alvimopan preoperatively.

  2. Subjects that have taken therapeutic doses of opioids for more than 7 days immediately prior to surgery.

  3. Subjects with severe hepatic impairment.

  4. Subjects with end-stage renal disease.

  5. Subjects who are pregnant.

  6. Subjects who have undergone imaging suggesting a small bowel obstruction.

  7. Subjects with a medical condition that may interfere with the use of the study medication Alvimopan.

  8. Subjects who have a condition or general disability or infirmity that in the opinion of the investigator precludes further participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Conor Delaney, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Story SK, Chamberlain RS. A comprehensive review of evidence-based strategies to prevent and treat postoperative ileus. Dig Surg. 2009;26(4):265-75. doi: 10.1159/000227765. Epub 2009 Jul 3. PMID 19590205
- [Background] Bauer AJ, Boeckxstaens GE. Mechanisms of postoperative ileus. Neurogastroenterol Motil. 2004 Oct;16 Suppl 2:54-60. doi: 10.1111/j.1743-3150.2004.00558.x. PMID 15357852
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Behm B, Stollman N. Postoperative ileus: etiologies and interventions. Clin Gastroenterol Hepatol. 2003 Mar;1(2):71-80. doi: 10.1053/cgh.2003.50012. PMID 15017498
- [Background] Luckey A, Livingston E, Tache Y. Mechanisms and treatment of postoperative ileus. Arch Surg. 2003 Feb;138(2):206-14. doi: 10.1001/archsurg.138.2.206. PMID 12578422
- [Background] Delaney CP, Brady K, Woconish D, Parmar SP, Champagne BJ. Towards optimizing perioperative colorectal care: outcomes for 1,000 consecutive laparoscopic colon procedures using enhanced recovery pathways. Am J Surg. 2012 Mar;203(3):353-5; discussion 355-6. doi: 10.1016/j.amjsurg.2011.09.017. Epub 2012 Jan 20. PMID 22264739
- [Background] Zhuang CL, Ye XZ, Zhang XD, Chen BC, Yu Z. Enhanced recovery after surgery programs versus traditional care for colorectal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2013 May;56(5):667-78. doi: 10.1097/DCR.0b013e3182812842. PMID 23575408
- [Background] Delaney CP, Wolff BG, Viscusi ER, Senagore AJ, Fort JG, Du W, Techner L, Wallin B. Alvimopan, for postoperative ileus following bowel resection: a pooled analysis of phase III studies. Ann Surg. 2007 Mar;245(3):355-63. doi: 10.1097/01.sla.0000232538.72458.93. PMID 17435541
- [Background] Delaney CP, Craver C, Gibbons MM, Rachfal AW, VandePol CJ, Cook SF, Poston SA, Calloway M, Techner L. Evaluation of clinical outcomes with alvimopan in clinical practice: a national matched-cohort study in patients undergoing bowel resection. Ann Surg. 2012 Apr;255(4):731-8. doi: 10.1097/SLA.0b013e31824a36cc. PMID 22388106
- [Background] Senagore AJ, Bauer JJ, Du W, Techner L. Alvimopan accelerates gastrointestinal recovery after bowel resection regardless of age, gender, race, or concomitant medication use. Surgery. 2007 Oct;142(4):478-86. doi: 10.1016/j.surg.2007.07.004. PMID 17950339
- [Background] Traut U, Brugger L, Kunz R, Pauli-Magnus C, Haug K, Bucher HC, Koller MT. Systemic prokinetic pharmacologic treatment for postoperative adynamic ileus following abdominal surgery in adults. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD004930. doi: 10.1002/14651858.CD004930.pub3. PMID 18254064
- [Background] Zingg U, Miskovic D, Pasternak I, Meyer P, Hamel CT, Metzger U. Effect of bisacodyl on postoperative bowel motility in elective colorectal surgery: a prospective, randomized trial. Int J Colorectal Dis. 2008 Dec;23(12):1175-83. doi: 10.1007/s00384-008-0536-7. Epub 2008 Jul 30. PMID 18665373
- [Background] Al-Mazrou AM, Baser O, Kiran RP. Alvimopan, Regardless of Ileus Risk, Significantly Impacts Ileus, Length of Stay, and Readmission After Intestinal Surgery. J Gastrointest Surg. 2018 Dec;22(12):2104-2116. doi: 10.1007/s11605-018-3846-2. Epub 2018 Jul 9. PMID 29987738
- [Background] Jang J, Kwok B, Zhong H, Xia Y, Grucela A, Bernstein M, Remzi F, Hudesman D, Chen J, Axelrad J, Chang S. Alvimopan for the Prevention of Postoperative Ileus in Inflammatory Bowel Disease Patients. Dig Dis Sci. 2020 Apr;65(4):1164-1171. doi: 10.1007/s10620-019-05839-5. Epub 2019 Sep 14. PMID 31522323
- [Background] Wen Y, Jabir MA, Keating M, Althans AR, Brady JT, Champagne BJ, Delaney CP, Steele SR. Alvimopan in the setting of colorectal resection with an ostomy: To use or not to use? Surg Endosc. 2017 Sep;31(9):3483-3488. doi: 10.1007/s00464-016-5373-0. Epub 2016 Dec 7. PMID 27928668
- [Background] Steele SR, Brady JT, Cao Z, Baumer DL, Robinson SB, Yang HK, Delaney CP. Evaluation of Healthcare Use and Clinical Outcomes of Alvimopan in Patients Undergoing Bowel Resection: A Propensity Score-Matched Analysis. Dis Colon Rectum. 2018 Dec;61(12):1418-1425. doi: 10.1097/DCR.0000000000001181. PMID 30312222
- [Background] Keller DS, Flores-Gonzalez JR, Ibarra S, Mahmood A, Haas EM. Is there value in alvimopan in minimally invasive colorectal surgery? Am J Surg. 2016 Nov;212(5):851-856. doi: 10.1016/j.amjsurg.2016.02.016. Epub 2016 May 10. PMID 27262754
- [Background] Hyde LZ, Kiely JM, Al-Mazrou A, Zhang H, Lee-Kong S, Kiran RP. Alvimopan Significantly Reduces Length of Stay and Costs Following Colorectal Resection and Ostomy Reversal Even Within an Enhanced Recovery Protocol. Dis Colon Rectum. 2019 Jun;62(6):755-761. doi: 10.1097/DCR.0000000000001354. PMID 30807457
- [Background] Asgeirsson T, El-Badawi KI, Mahmood A, Barletta J, Luchtefeld M, Senagore AJ. Postoperative ileus: it costs more than you expect. J Am Coll Surg. 2010 Feb;210(2):228-31. doi: 10.1016/j.jamcollsurg.2009.09.028. Epub 2009 Nov 18. PMID 20113944
- [Background] Iyer S, Saunders WB, Stemkowski S. Economic burden of postoperative ileus associated with colectomy in the United States. J Manag Care Pharm. 2009 Jul-Aug;15(6):485-94. doi: 10.18553/jmcp.2009.15.6.485. PMID 19610681
- [Background] Mao H, Milne TGE, O'Grady G, Vather R, Edlin R, Bissett I. Prolonged Postoperative Ileus Significantly Increases the Cost of Inpatient Stay for Patients Undergoing Elective Colorectal Surgery: Results of a Multivariate Analysis of Prospective Data at a Single Institution. Dis Colon Rectum. 2019 May;62(5):631-637. doi: 10.1097/DCR.0000000000001301. PMID 30543534
- [Background] Tevis SE, Carchman EH, Foley EF, Harms BA, Heise CP, Kennedy GD. Postoperative Ileus--More than Just Prolonged Length of Stay? J Gastrointest Surg. 2015 Sep;19(9):1684-90. doi: 10.1007/s11605-015-2877-1. Epub 2015 Jun 24. PMID 26105552

RESULTS

PARTICIPANT FLOW:
Groups:
- Alvimopan Group: Patients randomized to the study group will be given a maximum of 3 doses of Alvimopan 12mg orally, 12 hours apart. Alvimopan will be given from the time of diagnosis of postoperative ileus to the time of return of bowel function or the maximum 3 doses. Subsequent Alvimopan doses will be given if there is no return of bowel function or if symptoms of distension and/or nausea persist despite some return of bowel function.
  All patients will follow a standard ERAS pathway after surgery, with early feeding and ambulation, along with opioid minimizing measures as is our standard postoperative protocol.
  Alvimopan: Alvimopan will be given to patients who are diagnosed with postoperative ileus after surgery
Period: Overall Study
Arm/Group | Alvimopan Group | Control Group
Started | 33 | 32
Completed | 31 | 32
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Screen Failure- Received Alvimopan Preoperatively | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvimopan Group | Control Group | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 56 [43 to 66] | 63 [49 to 73] | 61 [46 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 21 | 20 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Number of days from postoperative ileus diagnosis until discharge from hospital
Time Frame: up to 30 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 31 | 32
days | 5 [3.5 to 6.5] | 6 [5 to 8]

2. Secondary Outcome: Time to Return of Bowel Function
Description: Number of days between Ileus diagnosis and time of passing flatus, stool and tolerating diet
Time Frame: up to 30 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 31 | 32
days | 1 [0 to 2] | 2 [1 to 3.5]

3. Secondary Outcome: Number of Participants With Re-operation
Description: Number of participants with re-operations within 30 days of surgery
Time Frame: within 30 days of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 31 | 32
Participants | 3 | 0

4. Secondary Outcome: Number of Participants With Re-admissions
Description: Number of participatnts with re-admissions within 30 days of surgery
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 31 | 32
Participants | 7 | 5

ADVERSE EVENTS:
Time Frame: 30 days following surgery
Arm/Group | Alvimopan Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 10/31 | 13/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvimopan Group (N=31) | Control Group (N=32)
Surgical Site Infection (Infections and infestations) | 0 (0) | 4 (4) — Surgical site infection Overall 4 (6.3%) Alvimopan 0 (0%) Control 4 (12.5%) P-value 0.11
urinary retention (Renal and urinary disorders) | 5 (5) | 6 (6) — Urinary retention overall 11 (17.5%) alvimopan 5 (16.1%) control 6 (18.8%) p-value 0.8
other post-op complication (General disorders) | 5 (5) | 3 (3) — Other post-op complications overall 8 (12.7%) alvimopan 5 (16.1%) control group 3 (9.4%) p-value 0.47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04405037/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT04405037/ICF_001.pdf